CLINICAL TRIAL: NCT06929117
Title: Prevalence of Types and Patterns of Gastrointestinal Polyps in Assiut University Hospitals ( Cross Sectional Study
Acronym: Polyp
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshimaa Ahmed Mohammed Nossier, Resident pathology doctor, Assiut University
Other Study IDs: Prevalence of GIT POlyps
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: GI Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal polyps (GIPs) are unusual growths of epithelial tissue projecting from the mucosa of gastrointestinal tract (GIT) and one of the most common pathologies affecting GIT . They are either proliferative or neoplastic mucosal lesions that are commonly seen in the colon and less commonly occur in the esophagus, stomach and small intestine. They may remain asymptomatic or present as bleeding, pain and obstruction due to mass effect. However, the most important risk with the gastrointestinal polyps is the development of malignancy in some of these polyps . Gastric polyps include hyperplastic, fundic gland polyps, inflammatory fibroid polyp, adenomas like pyloric gland adenoma, and oxyntic gland adenoma. Hyperplastic gastric polyps rarely undergo neoplastic progression (1.5-2.1%) but are associated with an increased risk of synchronous cancer occurring elsewhere in the gastric mucosa . Gastric adenomas are true neoplasms and precursors of gastric cancer. Adenomas larger than 20 mm in width and villous histology have a higher risk of neoplastic progression . The presence of gastric adenomas is strongly associated with synchronous or metachronous gastric adenocarcinoma . Polyps of the small bowel are rare compared to those of the colo-rectum, with adenomas being most common and having more preference for the distal duodenum, ampullary, and periampullary region Colonic Polyps may be classified according to their gross appearance (sessile or pedunculated), histopathological features (hyperplastic, adenoma, etc.), and behavior (benign or malignant). The biggest concern is their ability to progress into adenocarcinoma, through the adenoma to carcinoma sequence due to genetic mutation .

DETAILED DESCRIPTION:
Gastrointestinal polyps (GIPs) are unusual growths of epithelial tissue projecting from the mucosa of gastrointestinal tract (GIT) and one of the most common pathologies affecting GIT . They are either proliferative or neoplastic mucosal lesions that are commonly seen in the colon and less commonly occur in the esophagus, stomach and small intestine. They may remain asymptomatic or present as bleeding, pain and obstruction due to mass effect. However, the most important risk with the gastrointestinal polyps is the development of malignancy in some of these polyps . Gastric polyps include hyperplastic, fundic gland polyps, inflammatory fibroid polyp, adenomas like pyloric gland adenoma, and oxyntic gland adenoma. Hyperplastic gastric polyps rarely undergo neoplastic progression (1.5-2.1%) but are associated with an increased risk of synchronous cancer occurring elsewhere in the gastric mucosa . Gastric adenomas are true neoplasms and precursors of gastric cancer. Adenomas larger than 20 mm in width and villous histology have a higher risk of neoplastic progression . The presence of gastric adenomas is strongly associated with synchronous or metachronous gastric adenocarcinoma . Polyps of the small bowel are rare compared to those of the colo-rectum, with adenomas being most common and having more preference for the distal duodenum, ampullary, and periampullary region Colonic Polyps may be classified according to their gross appearance (sessile or pedunculated), histopathological features (hyperplastic, adenoma, etc.), and behavior (benign or malignant). The biggest concern is their ability to progress into adenocarcinoma, through the adenoma to carcinoma sequence due to genetic mutation . With the use of Colonoscopy as an outpatient procedure to see inside of the colon and rectum and used in screening, diagnostic and therapeutic of rectal and colon diseases It is vital to discover high-risk polyps during colonoscopy to prevent colorectal cancer. This necessitates a more comprehensive description including morphology, anatomical distribution, and histopathology of those precursor lesions within the entire colon. Among patients with sporadic colorectal polyps, it is important to identify those at risk for malignancy. According to histopathology, serrated polyps, small distal hyperplastic polyps (HPs) have no substantial malignant potential and do not affect colonoscopic surveillance intervals. However, sessile serrated lesions (SSL) and traditional serrated adenomas (TSA) increase the risk of colorectal carcinoma. Generally, high-risk adenoma refers to patients with 1 or more of the following findings: 3 or more adenomas, adenoma ≥10 mm in size, and adenoma with tubulovillous/villous or high-grade dysplasia (HGD) histology . Neoplastic polyps are accountable for roughly 5-10% of population over age of 40 and these are important predisposing factor for majority of large bowel carcinoma cases. The neoplastic polyps are of primary importance because they harbor a malignant potential, which represents a stage in the development of colorectal cancer. For this reason, it is essential to identify these polyps at a sufficiently early stage, when a simple procedure to remove them can stop the development of colorectal cancer and prevent disease and death .

Non neoplastic polyps are important differential diagnosis for the neoplastic polyps and they include: Hyperplastic polyps, Hamartomatous polyps (juvenile polyps) and inflammatory polyps (pseudopolyps). The histopathological study is essential to detect dysplasia.

ELIGIBILITY:
Inclusion Criteria:All patients diagnosed with Gastrointestinal polyp based on standard clinical, endoscopic, and histological criteria will be included in the study.

-

Exclusion Criteria:

* Patients with insufficient data were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This cross-sectional study will be conducted on all specimens with gastrointestinal polyps referred to the pathology Laboratories at ElRajhy hospital and surgical pathology lab in Assuit University Hospital during the period from January 2022 to December 2024 after approval of the committee of ethics of scientific research in Faculty of Medicine in Assuit University. The data will be collected from registers, medical files and reports from pathological department of Assiut University Hospital.Slides will be reviewed with Haematoxylin-Eosin stain to determinethe type of the polyps.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the presence and grade of dysplasia either low grade or high grade dysplasia in all examined polyps. | during the period from January 2022 to December 2024
  To assess the presence and grade of dysplasia either low grade or high grade dysplasia in all examined polyps.

REFERENCES:
- See also: D.Y. Park et al.Arch Pathol Lab Med(2008) — http://dx.doi.org/10.1053/s0887-7963(02)80145-6
- See also: Nomenclature Abstract for Fulvimonas Mergaert et al. 2002 — http://dx.doi.org/10.1601/nm.2236
- See also: Colitides: diagnostic challenges and a pattern based approach to differential diagnosis — http://dx.doi.org/10.1016/j.mpdhp.2017.11.001
- See also: Assarzadegan N, Montgomery E. Gastric polyps. Diagn Histopathol. 2017;23(12):521-9. — http://dx.doi.org/10.1007/s00428-018-2400-7